CLINICAL TRIAL: NCT04708938
Title: Effectiveness of Different Physiotherapy Practices in Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Halime ARIKAN, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 68869993-511.06-E.239934
Record Dates: First submitted 2021-01-10; First posted 2021-01-14 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Temporomandibular Disorder
Keywords: High voltage stimulation; Temporomandibular disorders; Temporomandibular joint; Cervical spine; Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, randomized-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): High voltage electrical stimulation + exercise therapy
  Interventions: Other: High voltage electrical stimulation+exercise therapy
- Control group (Active Comparator): Exercise therapy
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Other: High voltage electrical stimulation+exercise therapy — The effect of high voltage electrical stimulation on temporomandibular disorders
  Arms: Treatment group
Other: Exercise therapy — The effect of high voltage electrical stimulation on temporomandibular disorders
  Arms: Control group

SUMMARY:
The aim of the study is to examine the effect of high voltage electrical stimulation on pain, temporomandibular joint mobility, cervical mobility, head position, tender points and joint sounds in individuals with temporomandibular disorders.

DETAILED DESCRIPTION:
28 individuals who meet the TMER / Research Diagnostic Criteria classification will be randomly divided into 2 groups. Exercise with high voltage electrical stimulation (YVES) will be applied to the 1st group and only exercise will be applied to the 2nd group. The second group will be the control group of the study. Both groups will be informed about the disease before starting the study before the treatment and patient education will be given about the situations that need attention. Again, 2 groups will be given an exercise program from the day they start the treatment, 3 times a week for 4 weeks during the treatment. As sociodemographic information of the individuals, age, gender, height, weight, body mass index, marital and educational status, occupation, smoking and alcohol use, patient history, family history and complaint sides will be recorded. Before starting treatment, individuals will be evaluated for pain, temporomandibular joint mobility, cervical mobility, tender points, and joint sounds:

1. Pain with Visual Analogue Scale (VAS),
2. TMJ mobility with a ruler,
3. Cervical mobility with C-ROM (Cervical Range of Motion) inclinometer,
4. Head position with universal goniometer and ImageJ software,
5. Sensitive points with algometer,
6. Joint sounds will be evaluated as present / absent as a result of the evaluation of movements in all directions (maximum mouth opening, right / left lateral excursions, protrusion and retrusion).

After 4 weeks of treatment, the measurements will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have been diagnosed with TMER,
* Comply with the TMD / RDC classification,
* Have Class I-II-III occlusion,
* Volunteer to participate in the study, and fill out the informed consent form will be included.

Exclusion Criteria:

* Acute trauma,
* Surgery history,
* Neurological or psychiatric conditions,
* Trigeminal or postherpatic neuralgia,
* Dental or orofacial infection,
* Intraoral infection or tumor,
* Oligodontics and anadontics,
* High voltage electrical stimulation contraindications,
* Any disease diagnosed in the shoulder and neck areas,
* Receiving another treatment and,
* Individuals under the age of 18 will be excluded in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in pain on temporomandibular joint | Before and after treatment, 4 weeks apart. It takes 10 seconds.
  Pain with Visual Analogue Scale (VAS)
Change in temporomandibular joint mobility | Before and after treatment, 4 weeks apart. It takes 3 minutes.
  Temporomandibular joint mobility with a ruler
Change in cervical mobility | Before and after treatment, 4 weeks apart. It takes 5 minutes.
  Cervical mobility with C-ROM (Cervical Range of Motion) inclinometer
Change in head position | Before and after treatment, 4 weeks apart. It takes 3 minutes.
  Head position with universal goniometer and ImageJ software
Change in tender points | Before and after treatment, 4 weeks apart. It takes 10 minutes.
  Tender points with algometer
Change in joint sounds | Before and after treatment, 4 weeks apart. It takes 2 minutes.
  Joint sounds as present / absent as a result of the evaluation of movements in all directions (maximum mouth opening, right / left lateral excursions, protrusion and retrusion)

CONTACTS AND LOCATIONS:
Overall Officials: Halime ARIKAN, MSc., Principal Investigator — Gazi University, Faculty of Health Sciences; Gokhan MARAS, MSc., Principal Investigator — Gazi University, Faculty of Health Sciences; Seyit CITAKER, Dr., Principal Investigator — Gazi University, Faculty of Health Sciences; Cahit UCOK, Dr., Principal Investigator — Ankara University, Faculty of Dentistry
Locations (1):
- Gazi University, Faculty of Health Sciences, Ankara, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR